CLINICAL TRIAL: NCT05167071
Title: An Open-Label, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, PK/PD and Preliminary Efficacy of HBM4003 in Combination With Toripalimab/ Tislelizumab in Patients With Advanced NEN and Other Solid Tumors
Brief Title: HBM4003 Combine With Toripalimab in Patients With Advanced NEN and Other Solid Tumors Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4003.6
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors; Neuroendocrine Tumors; CRC
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — toripalimab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBM4003(dose 1) and Toripalimab (Experimental): Arm A: HBM4003(dose 1) combined with Toripalimab in patients with advanced NEN
  Interventions: Drug: HBM4003; Drug: Toripalimab
- HBM4003(dose 2) and Toripalimab (Experimental): Arm B: HBM4003(dose 2) combined with Toripalimab in patients with advanced NEN
  Interventions: Drug: HBM4003; Drug: Toripalimab
- HBM4003 and Tislelizumab (Experimental): Arm F: HBM4003(dose 1) combined with Tislelizumab in patients with advanced CRC
  Interventions: Drug: HBM4003; Drug: Tislelizumab

INTERVENTIONS:
Drug: HBM4003 — Subjects will be treated with HBM4003 on Day 1 during each 21-day cycle.
  Other Names: Porustobart
Drug: Toripalimab — Subjects will be treated with Toripalimab on Day 1 during each 21-day cycle.
  Arms: HBM4003(dose 1) and Toripalimab; HBM4003(dose 2) and Toripalimab
Drug: Tislelizumab — Subjects will be treated with Tislelizumab on Day 1 during each 21-day cycle.
  Arms: HBM4003 and Tislelizumab

SUMMARY:
To select RP2D/MTD of HBM4003 in combination with Toripalimab in dose confirmation part(Part 1) and use the RP2D in dose expansion part (Part 2) to evaluate the safety, tolerability, PK/PD and preliminary efficacy of in patients with advanced NEN and other solid tumors

DETAILED DESCRIPTION:
Subjects will be treated with HBM4003 in combination with Toripalimab for up to 2 years or until confirmed disease progression, unacceptable tolerability or treatment discontinuation through withdrawal of consent occurs, whichever happens first.

This trial consists of:

* A screening period: 28 days
* A treatment period: no longer than 2 years (Part 1 dose escalation study or Part 2 dose expansion)
* A post-treatment follow-up period, including 28 days and 84 days after the last dose of study drug;
* Survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years at the time of signing the informed consent form. For Part 1 of this study, the subjects should be ≤ 75 years of age.
2. Patients for Part 1: patients histopathologically diagnosed with advanced or recurrent solid tumors.
3. For arm A and B of Part 2 in the study, Patients with non- functional metastatic neuroendocrine tumor confirmed by histopathology.
4. For arm F of Part 2 in the study, Patients with metastatic colorectal adenocarcinoma diagnosed by histopathology.
5. Patients must be able to provide archived tumor tissues after latest treatment or fresh tumor tissues and relevant pathology report.
6. Patients whose estimated survival time is more than 3 months.
7. Patients with at least one measurable lesion at baseline according to RECIST (Version 1.1). The lesion had not previously received surgery, radiotherapy and/or local treatment.
8. Patients with Eastern Cooperative Oncology Group(ECOG) performance status score ≤1.
9. Every woman or man with potential fertility needs to use an effective contraceptive method during the study, up to within 3 months after last drug administration.
10. Willing and able to comply with study-specified visits schedule, treatment plan, laboratory examination and other study procedures.

Exclusion Criteria:

1. Patients who are simultaneously participating in another clinical study.
2. Patients with a history of severe allergic diseases, a history of severe drug allergies, and known or suspected allergy to macromolecular protein preparations or HBM4003 or Toripalimab or Tislelizumab or its excipients.
3. Previous and concomitant drugs or treatments to be excluded like:

   * Anti-CTLA4 drug;
   * For part 1, anti-PD1 anti-PDL1 or anti-PDL2 treatment was received within 8 weeks prior to the start of the study;
   * For part 2, patients received anti-PD1, anti-PDL1 or anti-PDL2 treatment during the relapse or metastasis stage, and the time from the last treatment is short than 12 months before the first dose;
   * Received other antitumor treatment (including chemotherapy, radiation, targeted therapy, or biotherapy), antitumor vaccine, chinese herbal medicine or proprietary medicine with anti-tumor effect, Immunosuppressant or glucocorticoid, Transfusion of PLT or RBC prior to initiation of study treatment;
   * live attenuated vaccine was received before study administration or planned during the study period.
4. Insufficient recovery from previous treatments.
5. Diseases that may affect the efficacy and safety of the investigational product, including but not limited to active infection, active autoimmune disease or autoimmune disease, primary immunodeficiency disease, any clinically significant cardiovascular disease, severe pulmonary insufficiency, organ transplantation, etc.
6. A history of other malignant diseases within 5 years before the first dose.
7. Symptomatic, active, or urgent treatment-requiring central nervous system (CNS) metastasis with imaging evidence (based on CT or MRI assessment).
8. Subjects with pleural effusion, pericardial effusion, or ascites that could not be stabilized by repeated drainage or other methods were determined by investigator.
9. Patients who the investigator believes may have other factors that will affect the efficacy or safety evaluation of this study (e.g., mental disorders, alcoholism, drug use, etc.).
10. Women who are pregnant or breastfeeding, or who plan to become pregnant during the study period and within 3 months after the last administration of the investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: DLT | approximate 21 days
  Number of subjects with DLT in each dose cohort within 1 cycle (21 days) after the first drug administration
Part 1: MTD | approximate 21 days
  The maximum tolerated dose (MTD) of HBM4003 combined with Toripalimab
Part 1: RP2D | approximate 21 days
  The recommended phase 2 dose (RP2D) of HBM4003 combined with Toripalimab
Part 2: ORR | maximum 2 years
  Proportion of subjects with complete response (CR) and partial response (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang P, Chen K, Yang J, Song L, Zheng F, Luo R, He Y, Li F, Yang D, Cao N, Tao X, Shen L, Lu M. Efficacy and safety of HBM4003 combined with toripalimab in refractory neuroendocrine neoplasms: a multicenter, phase II study. EClinicalMedicine. 2025 Jun 3;84:103249. doi: 10.1016/j.eclinm.2025.103249. eCollection 2025 Jun. PMID 40521168

DOCUMENTS (1):
  • Study Protocol (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05167071/Prot_001.pdf